CLINICAL TRIAL: NCT05002062
Title: The Influence of Cognitive Behavioral Therapy on Fatigue, Cognition and Inflammatory Biomarkers in Multiple Sclerosis Patients
Brief Title: Efficacy of Cognitive Behavioral Therapy on Fatigue, Cognition and Inflammatory Biomarkers in MS Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Engy Badreldin Saleh Moustafa, PhD, Lecturer of P.T for neuromuscular disorders and its surgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003199
Record Dates: First submitted 2021-06-12; First posted 2021-08-12 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: A Single Blinded, Randomized Controlled Trial
Who Masked: Participant
Masking Description: Sealed Envelopes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- G1 ( Conventional Physical Therapy Program group) (Sham Comparator): Patients in G1 underwent conventional physical therapy program continued for 3 months, included (aerobic training 20 minutes, resistive training for 15 minutes and flexibility program for 15 minutes).
  The whole treatment session lasted from 50 minutes to one hour, 3 times per week for 3 consecutive months.
  Interventions: Other: Conventional physical therapy program
- G2 ( Computer-based Cognitive Therapy group) (Active Comparator): Patients in G2 underwent Computer-based cognitive training continued for 3 months, included (attention/concentration, memory and reaction behavior training).
  The whole treatment session timing lasted 50 minutes to one hour, 3 times per week for 3 consecutive months.
  Interventions: Device: "RehaCom" computer-based cognitive training in addition to Conventional physical therapy program; Other: Conventional physical therapy program

INTERVENTIONS:
Device: "RehaCom" computer-based cognitive training in addition to Conventional physical therapy program — Rehacom procedure: It is a computer-based intensive cognitive rehabilitation test used to assess patient's cognitive functions. It includes 32 assessment tasks for attention, memory , logical reasoning& executive functioning. It composes of regular PC , 1G RAM , DVD drive, 100 GB hard drive with windows XP SP3, 128 MB RAM direct 3D graphic card , Screen at least 19" , regular PC keyboard or Rehacom panel & printer .The Rehacom software version is (patient enpult (1990-1997) EN/ISO-13485-certified). It is characterized by easy handling, close to reality , motivating for patients.
  Arms: G2 ( Computer-based Cognitive Therapy group)
Other: Conventional physical therapy program — Conventional physical therapy program for MS patients include aerobic training, resistive training and flexibility program

SUMMARY:
There is a rising concern about quality of life of multiple sclerosis (MS) patients has emerged. Cognitive dysfunction with primary fatigue and there correlation to the level of disease inflammatory process has got great interest in MS research .

The aim of the present study was to examine the influence of using a computer-based cognitive behavioral therapy on primary fatigue, cognitive dysfunction, and inflammatory biomarkers for patients with MS.

Patients and methods A total of 40 MS patients (Expanded Disability Status Scale<5) were divided into two groups, both groups are suffering cognitive decline (using RehaCom software to assess attention/concentration, memory and reaction behavior) with primary fatigue according to the Fatigue Severity Scale (FSS>36). Patients with depression and sleep problems were excluded from the study. Patients in both groups have elevated serum levels of tumor necrosis factor-α (TNF-α) and interferon-γ (IFN-γ).

Patients in (G1) underwent conventional physical therapy program for MS including aerobic training, resistive training and a flexibility program, patients in (G2) underwent an intensive computer-based cognitive program for attention, concentration, memory and reaction behavior using the RehaCom software.

The conventional physical therapy interventions for both (G1) sustained for three months, 45 minutes to 1 hour, 3 times/week. The computer-based cognitive behavioral therapy for patients in (G2) was prescribed as following (45 minutes to 1 hour a session, 3 times/week for continues three months).

DETAILED DESCRIPTION:
This study was done to to examine the influence of using a computer-based cognitive behavioral therapy on primary fatigue, cognitive dysfunction, and inflammatory biomarkers for patients with MS. This study was conducted in the time period between December 2020 till May 2021.

1. Subjects Selection:

   Forty MS patients were selected from Neurology Department Faculty of Medicine, Cairo University out-patient clinic , Multiple Sclerosis Research Unit, Cairo University and from Faculty of Physical Therapy ,Cairo University out-patient clinic. The patients were diagnosed and referred from a neurologist. All the patients were referred from a neurologist as a clinically definite MS according to Mcdonald criteria. The diagnosis was confirmed by MRI. The patients were assigned into two equal groups (Conventional physical therapy program)(G1) & ( Computer-based cognitive behavioral therapy)(G2).
   * Inclusion criteria:

     * All types and representations of MS patients were included in this study. - The age of the patients ranged from 20-45 years. - All the patients subjected to a standard neurological examination before participating in the study( sensory, motor, coordination , balance, gait and fundus examination).
     * All the patients were free from any other neurological problems.
     * Multiple sclerosis patients were subdivided into two equal groups (Conventional physical therapy program)(G1) & ( Computer-based cognitive behavioral therapy)(G2).
     * All included patients for both groups complained from fatigue for more than three months with total score of FSS ≥ 36.
     * All included patients complained of a cognitive decline for more than three months ( including attention, concentration or memory problems according to the RehaCom scores)
     * All the patients were ambulatory with mild to moderate disability according to the expanded disability status scale (EDSS) ≤ 5(Ambulatory without aid or rest for 200 meters).
     * Serum levels of tumor necrosis factor-α (TNF-α) and interferon-γ (IFN-γ) were elevated in all recruited patients for both groups.
     * All the patients were medically stable with absent or mild hemiparetic, ataxic, sensory or motor manifestations.
     * The main complain for all patients in both groups is the sense of fatigue and varying degrees of cognitive dysfunction.
     * All recruited MS Patients kept on their medications as glucocorticoids, amantadine , betaferon , hypnotics and modafinil throughout the study.
     * All patients were educated .
   * Exclusion criteria:

   The patients were excluded when they met one of the following criteria:
   * Severe visual, verbal or acoustic impairments that may interfere with cognition testing,
   * Serious chronic illness that could interfere with or modify assessment or treatment outcomes.
   * Low leukocyte count & elevated ESR as this interfere with cytokine levels.
   * Secondary causes of fatigue including severe depression ( beck depression inventory (BDI ≥ 21) and sleep disturbance ( Epworth sleepiness scale (ESS ≥ 12)
   * Inability to complete questionnaires study outcome measure as in severe cognitive impairment and illiteracy.
   * Magnetic resonance imaging (MRI) of the brain showed plaques within the cingulate gyrus, insula , temporo-basal cortical areas or diffuse patchy frontal lesions as they usually complain from cognitive impairment independent of fatigue.
2. Instrumentations & Procedures :

   A. Assessment Interventions:

   • Fatigue severity scale (FSS) : It is valid and reliable scale used to assess fatigue severity in MS patients , and to distinguish fatigued MS patients from non fatigued MS patients(Armutlu et al,2007). It is self reported questionnaire consisted of nine sentences. A list of statements/questions is provided. These statements are related to the different aspects of fatigue and how it affects the body.

   Expanded Disability Status Scale (EDSS)was used to exclude patients with fatigue secondary to moderate to severe disability. It provides a total score on a scale that ranges from zero to ten. The first levels 1.0 to 4.5 indicate people with a high degree of ambulatory ability. The subsequent levels 5.0 to 9.5 indicate loss of ambulatory ability. Grade (Zero) indicate normal neurologic exam. Grade (Five) indicate the ability of the patient to ambulate without aid or rest for 200 meter but disability is severe enough to impair full daily activities. (Ten) indicate death due to MS.

   Beck depression inventory scale (BDI) was used to exclude patients suffering from fatigue secondary to depression. It composed of twenty one questions each with four possible responses ranging from "zero to three". Each question assess a specific symptom common among people with depression.

   Epworth Sleepiness Scale (ESS)was used to exclude the patients suffering from fatigue secondary to sleep disturbance. It assess daytime sleepiness in people with multiple sclerosis . It consists of eight questions regarding sleep in different physiological and psychological conditions in multiple sclerosis patients.

   Rehacom Software to assess cognitive function : It is a computer-based intensive cognitive rehabilitation test used to assess patient's cognitive functions. It includes 32 assessment tasks for attention, memory , logical reasoning& executive functioning. It composes of regular PC , 1G RAM , DVD drive, 100 GB hard drive with windows XP SP3, 128 MB RAM direct 3D graphic card , Screen at least 19" , regular PC keyboard or Rehacom panel & printer .The Rehacom software version is (patient enpult (1990-1997) EN/ISO-13485-certified). It is characterized by easy handling, close to reality , motivating for patients.

   Blood analysis: A blood sample was collected from each patient in both groups before and after the 4 months treatment intervention. Assessment of patients on immunomodulatory therapy was postponed 36 hours from the last dose. Serum blood samples were immediately stored on ice. TNF-α and IFN- γ were measured using The Quantikine Human TNF-alpha & IFN-gamma Immunoassay ELISA kit . It is a 3.5 or 4.5 hour solid phase ELISA designed to measure human TNF-alpha & IFN-gamma in cell culture supernates, serum, and plasma. It contains E. coli-derived recombinant human TNF-alpha, IFN-gamma and antibodies raised against this protein and antibodies raised against the recombinant factor. It has been shown to accurately quantities the recombinant factor (http://www.rndsystems.com/Products/DIF57&sta00c/aqQ).

   B. Treatment Interventions:
   * Conventional Physical Therapy Program for patients in (G1):

   Including (aerobic training 20 minutes, resistive training 15 minutes and flexibility program for 15 minutes), total conventional PT session timing (45 to one hour), 3 times /week for subsequent 3 months.
   * Computer- based Cognitive training using Rehacom Software in addition to Conventional Physical Therapy Program in (G2) :

   Cognitive training including the attention/concentration, memory and reaction behavior domains, The time of each cognitive training session(45 to one hour), 3 times /week for consecutive 3 months.
   * Each domain in the cognitive training tests consists of one hundred levels of difficulty . Each level has an average 22 subtests. The maximum period of the session was about (60 minutes) for each patient with five minutes rest in between each level.
   * In Rehacom cognitive training, each patient is trained according to his/her primary cognitive level, which is predetermined during the assessment stage of the study.
3. Data Analysis and Statistical Design:

   * All analyses were performed on SPSS for Windows version 22 (IBM Corp., Armonk, NY, USA).
   * At the baseline assessment, the mean values among the two groups were compared by one-way ANOVA for independent samples for continuous data or chi squared for categorical data.
   * The effects of the treatment pre-intervention and immediately post intervention were examined using the two factor ANOVA with factors 'time' (baseline, immediately post treatment intervention) on FSS ,RehaCom Cognitive domains' scores ( attention/concentration, memory & reaction behavior), and serum levels data of tumor necrosis factor-α (TNF-α) and interferon-γ (IFN-γ).
   * Data were expressed as mean ± standard deviation (SD), A p value less than 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* All types and representations of MS patients were included in this study. - The age of the patients ranged from 20-45 years. - All the patients subjected to a standard neurological examination before participating in the study( sensory, motor, coordination , balance, gait and fundus examination).
* All the patients were free from any other neurological problems.
* Multiple sclerosis patients were subdivided into two equal groups, (Conventional physical therapy program group)(G1) & Computer-based Cognitive training program (G2).
* All patients in both groups complained from fatigue for more than two months with total score of FSS ≥ 36.
* All patients in both groups complained from varying degrees of cognitive decline persisted for more than 3 months.
* All the patients were ambulatory with mild to moderate disability according to the expanded disability status scale (EDSS) ≤ 5(Ambulatory without aid or rest for 200 meters).
* Main complain for all patients is sense of fatigue with varying degrees of cognitive decline.
* All the patients were medically stable with absent or mild hemiparetic, ataxic, motor or sensory manifestations.
* All patients were educated .

Exclusion Criteria:

* Severe visual, verbal or acoustic impairments that may interfere with cognition testing,
* Serious chronic illness that could interfere with or modify assessment.
* Low leukocyte count & elevated ESR as this interfere with cytokine levels.
* Secondary causes of fatigue including severe depression ( beck depression inventory (BDI ≥ 21) and sleep disturbance ( Epworth sleepiness scale (ESS ≥ 12)
* Inability to complete questionnaires study outcome measure as in severe cognitive impairment and illiteracy.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2021-05-18 (Actual); Study Completion 2021-06-07 (Actual)

PRIMARY OUTCOMES:
Level of primary fatigue | Changes from baseline to pre-intervention, Changes from Pre-intervention to immediately post intervention
  Level of fatigue is assessed using the Fatigue severity scale (FSS) , It is valid and reliable scale used to assess fatigue severity in MS patients. It is self reported questionnaire consisted of nine sentences. A list of statements/questions is provided. These statements are related to the different aspects of fatigue and how it affects the body.Grading of the scale range from " one to seven". Grade (seven) indicate that the patient strongly agrees with a particular statement. Grade (one) indicate the patient strongly disagree to this particular statement (Debouverie et al., 2002). At the end of assessment , if the added total scores were above 36. This indicated that the patient suffer from MS-related fatigue.
Level of Attention/concentration | Changes from baseline to pre-intervention, Changes from Pre-intervention to immediately post intervention
  Rehacom software is used to assess pre and post treatment cognitive function domains including level of Attention/concentration. Higher scores of attention/concentration indicated better cognitive function and vice versa.
Figural Memory | Changes from baseline to pre-intervention, Changes from Pre-intervention to immediately post intervention
  Rehacom software is used to assess pre and post treatment cognitive function domains including figural memory. Higher scores of immediate figural memory indicated better cognitive function and vice versa.
Mental Reaction behavior | Changes from baseline to pre-intervention, Changes from Pre-intervention to immediately post intervention
  Rehacom software is used to assess pre and post treatment cognitive function domains including Mental Reaction behavior. Higher scores of mental reaction behavior indicated better cognitive function and vice versa.
Serum levels of Tumor Necrosis Factor-alpha (TNF-alpha) and Interferon-gamma(INF-gamma) | Changes from baseline to pre-intervention, Changes from Pre-intervention to immediately post intervention
  The Quantikine Human TNF-alpha & IFN-gamma Immunoassay ELISA kit . It is a 3.5 or 4.5 hour solid phase ELISA designed to measure human TNF-alpha & IFN-gamma in cell culture supernates, serum, and plasma. (TNF-alpha) and (INF-gamma) results are measured in pg/ml, elevated levels of circulating TNF-α & IFN-gamma indicate that the case is deteriorating or progressing.

CONTACTS AND LOCATIONS:
Overall Officials: Moshera H Darwish, PhD, Study Director — Cairo University
Locations (1):
- Faculty of physical therapy, Cairo University, Giza, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: No
Share title and main instrumentations & procedures only.

DOCUMENTS (1):
  • Informed Consent Form (2020-12-23): https://cdn.clinicaltrials.gov/large-docs/62/NCT05002062/ICF_002.pdf